CLINICAL TRIAL: NCT07398820
Title: Association of Sedentary Behavior and Physical Activity With Gut Transit Time and Its Effect on Gut Microbiota Inflammatory and Carcinogenic Potential
Brief Title: IMPACT OF SEDENTARY BEHAVIOR IN THE HOMEOSTASIS OF THE DIGESTIVE ECOSYSTEM
Status: Completed | Type: Observational
Sponsor: Clínica Universidad de los Andes (Other)
Collaborators: University of Chile (Other)
Responsible Party: Principal Investigator, Javiera Cancino Ramirez, Principal investigator, Clínica Universidad de los Andes
Other Study IDs: FAIN202201
Record Dates: First submitted 2024-11-07; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Colorectal Adenoma
Keywords: exercise; sedentary behavior; colorectal cancer; gut microbiota
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Individuals who have undergone a colonoscopy with a normal result.
  Interventions: Other: Initial assessment
- Polyps: Individuals who have undergone a colonoscopy with the result of colorectal adenoma
  Interventions: Other: Initial assessment

INTERVENTIONS:
Other: Initial assessment — Patients will be cited to the clinic for an initial assessment that will include:
  * Brief interview to identify health conditions and medicines
  * Fecal sample recollection for determination of gut microbiota composition
  * Physical activity assessment with 7-day accelerometry
  * Body composition through octopolar bioimpedance
  * Heart rate variability with a heart rate monitor
  * Food ingestion through a questionnaire

SUMMARY:
This study seeks to determine the relationship between sedentary behavior, gut transit, gut microbiota and polyps development. Will be conducted an evaluation which includes assessments of physical activity behaviors (through accelerometry), gut transit time (ingestion of two blue colored muffins), food ingestion (online nutritional survey), body composition (through bioimpedance), heart rate variability (with a heart rate monitor) and gut microbiota composition (from a fecal sample).

The main goal of this study is to see if there is a relationship between high sedentary time and a slower gut transit time, altering gut microbiota favoring dysbiosis and promoting polyps development. For this objective, it will be described gut microbiota composition (identifying which bacteria are present in the gut and in what quantities are they found), physical activity and sedentary behaviors time, gut transit time (how long does it take to defecate after eating a meal) in order to relate these factors with the presence of polyps.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* 40-60 years of age.
* Omnivorous diet.
* Negative or positive colonoscopy result with adenomatous polyp during the last 12 months.

Exclusion Criteria:

* Antibiotic treatment during the previous month.
* Daily use of aspirin.
* Chronic inflammatory bowel disease (Crohn's disease, ulcerative colitis).
* Chronic constipation or diarrheic syndrome.
* Autoimmune disease (such as celiac disease, type 1 diabetes, etc.).
* HIV.
* Food allergies.
* Chronic use of laxatives.
* Previous digestive surgery except appendicitis.
* Familial adenomatous polyposis or Lynch disease.
* Obesity (BMI>30) and/or type 2 diabetes mellitus.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients' recruitment will be conducted at Clínica Universidad de los Andes. Universe will include all subjects between 40-60 years of age who have undergone a colonoscopy during the previous year at Clínica Universidad de los Andes with a negative (control) or positive result with the presence of adenomatous polyp.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Gut microbiota composition | From enrollment to the end of the 7 days period of recollection.
  DNA will be extracted from fecal samples and will be sequenced by Illumina platform. After bioinformatics analysis, the alpha and beta diversity will be reported, as well as compositional data from single relevant taxa. Results will be expressed as relative abundance for each bacterial taxa.
Fecal metabolites | 7 days after enrollment
  Quantification of fecal short chain fatty acids (butyrate, propionate, acetate, valerate, isobutyrate and isovalerate) will be performed in a gas chromatograph. Concentration of other fecal metabolites derived from protein degradation will also be determined: ammonia by using a commercial kit; indole through colorimetry test; p-cresol and hydrogen sulfide will be identified using high performance liquid chromatography.
  Gut inflammation will be assessed through fecal calprotectin levels.

SECONDARY OUTCOMES:
Body composition | First day of enrollment
  Body composition will be assessed through octapolar bioimpedance. Individuals will have to stand barefoot in the scale and will be recorded:
  * Weight
  * Fat mass
  * Fat free mass
Food ingestion | 7 days from enrollment
  Dietary intake will be assessed with a Food Frequency Questionnaire designed and performed by a trained dietitian.
Gut transit time | From enrollment to the end of the 7 days period of recollection.
  Total gut transit time will be assessed through the blue dye method according to the protocol proposed by Asnicar et al. (2021). The subjects should eat two 'blue' muffins (84.5 g×2 with 0.75 g of Wilton 'royal blue' food coloring paste each) within a 10-minute period. For total gut transit time determination participants will be asked to register the day and hour of the first stool with blue dye along with their consistency based on Bristol scale. Bristol scale is a graded visual scale of stool type that gives a score from 1 (hard lumps) to 7 (watery diarrhea). Participants will have also a register sheet to write the day and hour of every spontaneous bowel movement during the week of use of the accelerometer. The register sheet must be returned to the investigator.
Psychological well-being | 7 days after enrollment
  Psychological well-being will be assessed through Ryff's Psychological Well-Being Scale . The shortened and validated Spanish version of Ryff's Scale will be used. The total score will be calculated by adding the scores for all question items. The higher the score, the better the psychological well-being is. The questionnaire will be sent to the subjects by e-mail.
Anxiety and depression | 7 days after enrollment
  Anxiety and depression will be assessed through Hospital Anxiety and Depression Scale (HADS). The Spanish version of HADS will be used which comprises 14 items divided into two subscales, anxiety and depression, each one with 7 items. The items are assessed through a Likert scale ranging from 0 to 3, with a score of 0 to 7 indicating no symptoms; a score of 8 to 10 indicating borderline case; and a score of 11 to 21 indicating clear symptoms of depression and/or anxiety. The questionnaire will be sent to the subjects by e-mail.
Physical activity and sedentary behavior | 7 days after enrollment
  Sedentary behavior will be assessed through accelerometry. The protocol for assessment and data analysis was adapted following the recommendations of Migueles et al. (2017). Accelerometers will be programmed to record at a frequency sampling of 90 Hz with a normal filter and with a time-sampling interval (epoch) every 60 seconds. Every subject should wear the accelerometer (wGT3X-BT, Actigraph) on their hip for 7 consecutive days during the 24 hours, except for water activities (shower and/or swimming). Non-wear-time will be defined as every period of more than 60 consecutive minutes with 0 counts per minute (cpm) and without interruptions. Every day with a wear-time of at least 16 hours will be considered as a valid day. Data will be considered valid when contain a record of at least four valid days including at least one day of the weekend. The acceleration and time spend in light, moderate and vigorous physical activity, as well as in sedentary behaviors will be reported.
Heart rate variability | First day of enrollment
  Heart rate variability will be assessed with a polar H9 monitor worn in the chest for a 5 minutes period. Spectral analysis of the RR segments will be interpreted as follows: high frequency peak (HF; 0.15-0.4 Hz) representing primarily parasympathetic modulation, low frequency peak (LF; 0.04-0.15 Hz) reflecting both sympathetic and parasympathetic modulation. LF and HF power will be calculated in milliseconds2 (ms2). The LF/HF ratio will be used as a marker of the relative degree of sympathetic-cardiac modulation. Total power (ms2) was used as an indicator of the overall variability of the RR intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Universidad de los Andes, Las Condes, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Gut microbiota FASTQ files along with the metadata will be upload to the open data repository Zenodo.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after publication
Access Criteria: The FASTQ files will be available in the open repository ZENODO with the relevant metadata. Any other information can be requested by email supported by a proposal that should describe planned analyses.